CLINICAL TRIAL: NCT05557734
Title: Comparative Study Between Caudal and Perianal Block on Intraoperative Anal Sphincter Muscle Tone and Postoperative Analgesia During Anal Sphincter Sparing Procedures Under General Anesthesia
Brief Title: Compartive Study Between Caudal and Perianal Block During Anal Sphincter Sparing Procedures Under General Anesthesia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Abd elmoneim Adel Abd elmoneim, clinical professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: MD-276-2021
Record Dates: First submitted 2022-09-24; First posted 2022-09-28 (Actual); Last update posted 2023-12-21 (Actual); Status verified 2023-12

CONDITIONS: Acute Post Operative Pain; Motor Activity
Keywords: caudal; perianal block; anal sphincter sparing procedures; postoperative pain
MeSH Terms: conditions — Pain, Postoperative; Motor Activity

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Masking Description: Double blinded(the surgeon and the outcome assessor)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- caudal epidural group (Active Comparator): the patient will be positioned in lateral position, sterilized from the iliac crest margin to the lower buttock by betadine and will be covered by sterile drapes exposing the sacral area. Sacral horns will be palpated and sacral hiatus and epidural area will be determined at S4-S5 level through the ultrasound. Short axis (transverse) will be used first to identify the two sacral cornua as two hyperechoic reverse U-shaped structure "Frog sign" and the sacrococcygeal ligament in between and epidural space beneath. An 18-gauge epidural needle (length 90 mm) will be used for direct puncture of sacrococcygeal membrane out of plane then the probe will be rotated to long axis (longitudinal) and the needle will be seen in plane in the epidural space. Injection of 40 ml 0.125% bupivacaine will expand the epidural space. The patient will be repositioned to lithotomy position and surgery will start after 5 min. of preparing the patient and sterilization to the surgery
  Interventions: Procedure: caudal block
- perianal block group (Active Comparator): , the patient will be in the lithotomy position, paint and drape the area of the block under strict aseptic precaution, draw a circle with a radius of 2.5cm around anal opening, mark a point at 2,4,8,10 clock position, prepare 40 ml 0.125% bupivacaine, use 1.5-inch 23/24 gauge needle connected to 10 ml syringe, insert full length of the needle into the ischiorectal fat immediately peripheral to the external sphinchter. This injection scheme target the terminal nerve branches of the anus rather than blocking the trunk of major nerves. At 2 clock position, inject 2-3 ml of LA with tilting in lateral direction,withdraw needle 1cm and after every 1cm inject 2-3ml of LA, repeat procedure at 4,8,10 clock position, remaining around 10 ml of LA is used to infiltrate in subcutaneous tissue in circumference of anal opening.
  Interventions: Procedure: perianal block

INTERVENTIONS:
Procedure: caudal block — injection of local anesthestic through the scral hiatus into the sacral canal to reach caudal epidural space
  Other Names: caudal epidural block
  Arms: caudal epidural group
Procedure: perianal block — local anesthestic infiltration in the perianal area to block terminal branches of the nerves supplying the anal canal
  Arms: perianal block group

SUMMARY:
Anal fistula is an abnormal tract communicating an external opening in the perianal skin with an internal opening in the anal canal. Anal fistula is treated by fistulotomy . sphincter sparing procedures are usually done under general anesthesia omitting neuromuscular blocking agents in order to preserve sphincter tone intraoperatively. The aim of this study is to evaluate the effect of caudal block analgesia versus perianal block analgesia combined with general anesthesia on the postoperative analgesic profile and the tone of external anal sphincter in sphincter sparing surgery.

DETAILED DESCRIPTION:
Anal fistula is an abnormal tract communicating an external opening in the perianal skin with an internal opening in the anal canal. Anal fistula is treated by fistulotomy . sphincter sparing procedures are usually done under general anesthesia omitting neuromuscular blocking agents in order to preserve sphincter tone intraoperatively.

The study will be designed to recruit 46 patients who have complex anal fistula and will be scheduled for sphincter sparing surgery.

All patients will receive routine preanesthetic evaluation. They will be kept fasting for2 hours for clear fluids and at least 8 hours for solid food prior to performing the block. On arrival in the operating room, heart rate (HR), non invasive blood pressure, oxygen saturation (SPO2) and electrocardiography monitors will be applied and the baseline values will be noted. Intravenous access (IV) will be secured and an appropriate IV fluid will be started.

Patients will receive general anesthesia with induction of 2mg/kg IV propofol, 1mcg/kg IV fentanyl and laryngeal mask insertion in supine positionand maintenance of anesthesia with isoflurane inhalation.

Patients will be randomly allocated into two study groups;

* 1st group (caudal block group): will receive general anesthesia with ultra sound (u/s) guided caudal block with 40 ml 0.125% bupivacaine (10 ml bupivacaine + 30 ml normal saline 0.9%).
* 2nd group (perianal block group): will receive general anesthesia with perianal block analgesia with 40 ml 0.125% bupivacaine (10 ml bupivacaine + 30 ml normal saline 0.9%).

Intraoperative, optimal surgical conditions and persistence of muscle tone will be determined by the general surgeon according to patient's anal sphincter relaxation using Digital Rectal Examination Scoring System (DRESS) which ranges from 0 to 5 but with usage of resting pressure only without squeezing pressure as the patient is anesthetized.

Postoperativepain control regimen will be used for the two groups as Paracetamol 15mg/kg IV /6 hours, Ketorlac 30 mg IV /8hours. A rescue analgesic dose of opioid in the form ofMorphine 0.05mg/kg as needed on patient demand if numeric pain score is more than three to be repeated every 20 min. till maximum dose 0.2mg/kg. if numerical rating score persists more than three.

ELIGIBILITY:
Inclusion Criteria:

* 18-60 years old patients
* ASA I-IIIpatients
* Patients with complex anal fistula

Exclusion Criteria:

* known hypersensitivity to amide type local anesthetics
* Patients with contraindications to caudal block or perianal block: use of anticoagulant medication, local infection in the intervention site, increased intracranial pressure and severe aortic and / or mitral valve stenosis.
* Patients who do not accept regional anesthesia
* BMI (Body mass index) > 35 kg/m2
* Anatomical abnormalities and previous surgeries involving the sacrum

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2023-10-14 (Actual); Primary Completion 2024-01 (Estimated); Study Completion 2024-02 (Estimated)

PRIMARY OUTCOMES:
time to first analgesic request after the recovery of the patient. | 24 hours
  duration of postoperative analgesia

SECONDARY OUTCOMES:
postoperative pain intensity | 24 hours
  pain measurement will be done using 11 point Numerical rating scale (0-10).
Assessment of External anal sphincter muscle tone intraoperative | 2 hours
  Digital Rectal Examination Score System(DRESS) 0 no descernable tone at rest
  1. very low tone
  2. mildly decreased tone
  3. Normal
  4. Elevated Tone
  5. Very high tone, atight anal canal
Total post operative opioid consumption | 24 hours
  total amount of morphine consumed by the patient in the postoperative period
incidence of complications | 24 hours
  bradycardia,Hypotension, postoperative nausea and vomiting,urine retention

CONTACTS AND LOCATIONS:
Overall Officials: Osama M Assad, professor, Principal Investigator — Anesthesia department , cairo university; Amany H Saleh, assprofessor, Study Director — Anesthesia department , Cairo university; Mona H Elsherbiny, lecturer, Study Chair — Anesthesia department , cairo university
Locations (1):
- Cairo university hospitals, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No